CLINICAL TRIAL: NCT07321691
Title: Evaluation of the Effectiveness of a Rehabilitation Program for Hearing and Communication Disorders in Elderly People in Nursing Homes: a Single Case Experimental Design (N of 1 Trials Study)
Brief Title: Evaluation of the Effectiveness of a Rehabilitation Program for Hearing and Communication Disorders in Elderly People in Nursing Homes.
Acronym: HEAR2SHARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/23/0390; 2025-A01543-46 (Other: ID-RCB)
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Deafness
Keywords: deafness; rehabilitation; nursing homes; elderly subject
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design (SCED) consists in repeated measures in a small sample size. Each subject acts as his own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- transmitter with receiver (Experimental): hearing rehabilitations : a transmitter with several receivers
  Interventions: Other: use of hearing rehabilitation device
- listening assistant. (Active Comparator): one type of hearing rehabilitations
  Interventions: Other: use of hearing rehabilitation device
- No hearing device (No Intervention): no hearing device

INTERVENTIONS:
Other: use of hearing rehabilitation device — the use hearing rehabilitation devices aimed to improve audibility
  Arms: listening assistant.; transmitter with receiver

SUMMARY:
In France, 64% of residents in nursing homes have moderate to severe hearing loss and only 12% are treated with hearing aids. Yet the extra-auditory consequences of presbycusis are numerous: general fatigue, isolation, anxiety and depression. France counted 620 000 nursing home beds in 2020 and this number increases each year by an average of 2% (DREES (Department of Research, Studies, Evaluation and Statistics), France, 2019). Only few studies have focused on hearing disorders in this population, given the importance of their communication difficulties (Solheim J et al., 2016, Kimball A et al., 2017 ). The population in nursing homes is for 80% over 80 years old (DREES (Department of Research, Studies, Evaluation and Statistics) survey, France, 2014). This same survey looked at the proportion of people with functional hearing limitations and their severity depending on where they live. The highest rates were found among people living in institutions (regardless of the degree of functional hearing limitations), with 42% of people living in nursing homes and senior residences who have hearing functional limitations against 15.9 % of those living at home The present study is interested in the management of hearing and communication disorders in nursing homes residents by setting up a program for the rehabilitation of these disorders, based on the use of a simple hearing device by the nursing home staff.

DETAILED DESCRIPTION:
The main objective of this study is to assess the effectiveness of a rehabilitation program for hearing and communication disorders intended to improve the communication of residents in nursing homes.

This program includes for the resident:

* the alternative use of two hearing rehabilitation devices aimed to improve audibility
* An inaugural training led by a trained professional to promote oral communication The effectiveness of the two devices will be compared.

This program includes for the staff members:

- A one-day training comprising three components (general concepts concerning deafness and its rehabilitation, training in the use of the device to improve audibility, training in facilitating the communication workshop).

ELIGIBILITY:
Inclusion Criteria:

* residents in nursing homes with hearing impairment (HHIE-S (Hearing Handicap Inventory for the Elderly Screening and pure tone audiometry)
* with an MMS (Mini Mental State) score> 15
* with a GIR Group ≥ à 3 affiliated to a social security scheme
* French speaking

Exclusion Criteria:

* wearing any type of hearing aid at the time of inclusion

  * having followed a similar training program
  * Subjects under juridical protections or tutelage measure
  * unable to answer questions and participate in group activities
  * with associated life-threatening pathologies and/or a life expectancy in EHPAD of less than 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
effectiveness of the Hear2Share program | every weeks from enrollment until end of participation at 15 weeks
  The primary outcome will be the effectiveness of the Hear2Share program evaluated by the Percentage of words correctly identified at 60 dB HL measured every weeks

SECONDARY OUTCOMES:
wearing time of the device | From enrollment to the end of participation at 15 weeks
  wearing time of the device in hours and every weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No